CLINICAL TRIAL: NCT07169916
Title: Effect of Yueju Pill Combined With Standard Therapy on Quality of Life and Treatment Efficacy in Patients With Advanced Biliary Tract Cancer: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Yueju Pill Combined With Standard Therapy In Advanced Biliary Tract Cancer
Acronym: YJ-BTC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Geriatric Medical Center (Other); Minhang Central Hospital (Unknown); Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Principal Investigator, Jia Fan, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YJ-BTC Trial
Record Dates: First submitted 2025-08-21; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Cancer (BTC)
Keywords: Biliary Tract Cancer; Yueju Pill; Quality of Life; Treatment Efficacy
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. Subjects, investigators, site staff, CRCs, and assessors will remain blinded to the intervention (Yueju Pill or placebo). Study drug and placebo are identical in appearance, packaging, color, odor, specifications, and labeling. Standard-of-care treatment is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yueju group (Group A) (Experimental): In addition to guideline-based standard therapy, patients will receive Yueju Pill according to the instructions, 6-9 g per dose, twice daily, orally, continued until tumor progression or until the patient is unable to continue treatment for other reasons.
  Interventions: Drug: Yueju Pill + Standard Anti-tumor Therapy
- Placebo group (Group A) (Placebo Comparator): Patients will receive guideline-based standard therapy combined with a placebo. The placebo is matched to Yueju Pill in appearance, smell, packaging, administration method, dosage, and treatment schedule.
  Interventions: Drug: Placebo + Standard anti-tumor therapy

INTERVENTIONS:
Drug: Yueju Pill + Standard Anti-tumor Therapy — Group A (Intervention): Standard therapy + Yueju Pill (6-9 g per dose, twice daily, orally until disease progression or intolerable toxicity).
  Arms: Yueju group (Group A)
Drug: Placebo + Standard anti-tumor therapy — Group B (Control): Standard therapy + placebo (identical in appearance, packaging, dosage, and administration frequency to Yueju Pill).
  Arms: Placebo group (Group A)

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the impact of Yueju Pill on quality of life and treatment efficacy in patients with advanced biliary tract cancer (BTC) receiving standard therapy.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled clinical trial aims to evaluate the impact of Yueju Pill on quality of life and treatment efficacy in patients with unresectable advanced or metastatic biliary tract cancer (BTC) receiving guideline-based standard chemotherapy. The study will be conducted at Zhongshan Hospital Affiliated with Fudan University, Xuhui District Central Hospital of Shanghai, Minhang District Central Hospital of Shanghai, and Shanghai Geriatric Medical Center. Eligible patients will be randomized into two groups: Group A (Intervention): Standard chemotherapy + Yueju Pill (6-9 g per dose, twice daily, orally until disease progression or intolerable toxicity). Group B (Control): Standard chemotherapy + placebo (identical in appearance, packaging, dosage, and administration frequency to Yueju Pill).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in this study:

1. No gender restriction, age ≥18 years, and expected survival ≥3 months;
2. ECOG Performance Status (PS) of 0-1;
3. Child-Pugh class A;
4. Histologically confirmed diagnosis of advanced biliary tract cancer (BTC), including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, or gallbladder cancer;
5. At least one measurable lesion according to RECIST v1.1 criteria;
6. Planned to receive or currently receiving guideline-based, chemotherapy-centered systemic first- or second-line therapy;
7. Presence of mild to moderate anxiety or depressive symptoms (PHQ-9 or GAD-7 score of 5-14);
8. Adequate major organ function, including:

   1. Hematology (no blood transfusion or hematopoietic growth factors within 14 days): Hb ≥90 g/L, ANC ≥1.5×10⁹/L, PLT ≥90×10⁹/L, WBC ≥3.0×10⁹/L;
   2. Biochemistry: TBIL ≤1.5×ULN (≤2×ULN if liver metastases); ALT and AST ≤2.5×ULN (≤5×ULN if liver metastases); serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min; plasma albumin ≥30 g/L;
   3. Coagulation: INR and PT ≤1.5×ULN, APTT ≤1.5×ULN;
   4. Cardiac function: LVEF ≥50%, QTcF ≤450 msec (male) or ≤470 msec (female);
   5. Urine protein ≤2+, and if >2+, 24-hour urine protein must be ≤1.0 g;
9. Not pregnant or breastfeeding, and subjects of childbearing potential must use effective contraception during treatment and for 3 months after treatment;
10. Voluntary participation with signed informed consent, good compliance, and willingness to cooperate with follow-up.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be eligible for this study:

1. Histological types of ampullary cancer, hepatocellular carcinoma, mixed-type liver cancer, or other malignancies not originating from bile duct cells;
2. History of or concurrent malignancy at other sites;
3. Severe anxiety or depression (PHQ-9 or GAD-7 score ≥15), currently receiving antidepressant or anti-anxiety medication, or history of substance abuse, alcoholism, or drug abuse;
4. Currently using other traditional Chinese medicine compound interventions;
5. Known allergy to monoclonal antibodies, anti-angiogenic drugs, gemcitabine, platinum drugs, or components of Chinese medicine;
6. Uncontrolled severe comorbidities, including:

   1. Congestive heart failure;
   2. Difficult-to-control hypertension;
   3. Angina or arrhythmias;
   4. Interstitial lung disease or active pulmonary tuberculosis;
   5. HBV DNA >2000 copies/mL or HCV RNA >1000 IU/mL after antiviral therapy;
   6. Known HIV positive or diagnosed with acquired immunodeficiency syndrome (AIDS);
   7. Clinically significant gastroesophageal variceal bleeding within 3 months prior to enrollment, or known bleeding tendency;
   8. Coagulation abnormalities (PT >14 sec), bleeding tendency, or currently receiving anticoagulant/thrombolytic therapy;
   9. Known or suspected active autoimmune disease, or requiring long-term systemic immunosuppressive therapy or corticosteroids;
7. Other factors that, in the investigator's judgment, may affect patient safety or trial compliance (e.g., severe laboratory abnormalities, psychiatric disorders, lack of family or social support).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in quality of life | 18 week after treatment
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 v3) was used to assess changes (Δ) in quality-of-life scores from baseline to week 18 after treatment. Scores on the EORTC QLQ-C30 range from 0 to 100, with higher scores indicating better global health status/quality of life.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score | 1 year
  The EORTC QLQ-C30 is a 30-item validated instrument assessing cancer-related quality of life across domains including physical, role, emotional, cognitive, and social functioning. Scores are transformed to a 0-100 scale. For functional and global health/QoL scales, higher scores indicate better quality of life. For symptom scales, higher scores indicate worse symptoms.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Cholangiocarcinoma Module (EORTC QLQ-BIL21) Score | 1 year
  The EORTC QLQ-BIL21 is a 21-item validated module designed for patients with cholangiocarcinoma, assessing disease-related symptoms and impact. Scores are transformed to a 0-100 scale, with higher scores indicating worse symptoms.
Objective response rate (ORR) | 1 year
  defined according to RECIST v1.1 criteria, calculated as the proportion of patients achieving complete response (CR) or partial response (PR) among all evaluable patients (CR + PR).
Disease control rate (DCR) | 1 year
  defined according to RECIST v1.1 criteria, calculated as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) among all evaluable patients (CR + PR + SD).
Overall survival (OS) | 1 year
  defined as the time from randomization to death from any cause or to the date of the last follow-up, whichever occurs first.
Progression-free survival (PFS) | 1 year
  defined as the time from randomization to the first documented disease progression by imaging or death from any cause, whichever occurs first.
Patient Health Questionnaire-9 (PHQ-9) Score | 1 year
  The Patient Health Questionnaire-9 is a 9-item self-report instrument measuring depressive symptoms. Scores range from 0 (no depressive symptoms) to 27 (severe depression). Higher scores indicate worse depressive symptoms.
Generalized Anxiety Disorder-7 (GAD-7) Score | 1 year
  The Generalized Anxiety Disorder-7 is a 7-item self-report instrument measuring anxiety symptoms. Scores range from 0 (no anxiety symptoms) to 21 (severe anxiety). Higher scores indicate worse anxiety symptoms.
Change in Traditional Chinese Medicine (TCM) syndrome score | 1 year
  the study-specific TCM Syndrome Information Scale will be used to assess changes and improvement in patients' TCM syndrome characteristics before and after treatment. Scores range from 0 to 100, with higher scores indicating more severe TCM symptoms (worse outcome).

OTHER OUTCOMES:
Incidence of treatment-related adverse events (AE/SAE) | 1 year
  all adverse events will be recorded and graded according to the NCI CTCAE v5.0 criteria, including but not limited to nausea, vomiting, and hepatic function abnormalities, with frequency and severity summarized.
Serum Cortisol Concentration | Baseline and at the end of each treatment cycle (each cycle is 21 days) during the treatment period.
  Cortisol levels in peripheral blood will be measured as a biomarker of stress response. Concentrations will be quantified using immunoassay.Unit of Measure: μg/dL
Serum Amino Acid Concentrations | Baseline and at the end of each treatment cycle (each cycle is 21 days) during the treatment period.
  Peripheral blood levels of selected amino acids (e.g., tryptophan, glutamine, arginine) will be measured as metabolic biomarkers using liquid chromatography-mass spectrometry (LC-MS).Unit of Measure: μmol/L
Composite Distribution of Peripheral Immune Cell Subsets | Baseline and at the end of each treatment cycle (each cycle is 21 days) during the treatment period.
  The proportion of major immune cell subsets in peripheral blood will be assessed by flow cytometry. The composite outcome includes:
  T lymphocytes (CD3+) CD4+ T cells (CD3+CD4+) CD8+ T cells (CD3+CD8+) B lymphocytes (CD19+ or CD20+) Natural killer (NK) cells (CD3-CD56+ and/or CD16+CD56+) Each component will be reported as the percentage of peripheral blood mononuclear cells (PBMCs). The composite outcome is defined as the 5-component vector of these percentages, with summary statistics (mean, SD, median, IQR) and changes from baseline presented for each subset.Unit of Measure: % of PBMCs
Inflammatory Cytokine Panel Score | Baseline and at the end of each treatment cycle (each cycle is 21 days) during the treatment period.
  A composite score reflecting systemic inflammatory cytokine burden will be calculated from serum/plasma concentrations of tumor necrosis factor-alpha (TNF-α), interleukin-6 (IL-6), interleukin-1β (IL-1β), interleukin-2 receptor (IL-2R), interleukin-8 (IL-8), and interleukin-10 (IL-10). For each cytokine, values will be standardized as z-scores relative to the study population, and the panel score will be defined as the sum of these standardized values. Higher scores indicate a higher overall inflammatory cytokine burden.
Serum Epinephrine/Norepinephrine Concentration | 1 year
  Epinephrine/Norepinephrine levels in peripheral blood will be measured as a stress-related catecholamine biomarker. Concentrations will be quantified using immunoassay.Unit of Measure: pg/mL
Serum Serotonin (5-HT) Concentration | Baseline and at the end of each treatment cycle (each cycle is 21 days) during the treatment period.
  Peripheral blood serotonin (5-HT) levels will be measured as a neurotransmitter biomarker. Concentrations will be quantified using immunoassay or high-performance liquid chromatography (HPLC).Unit of Measure: ng/mL
Serum Gamma-Aminobutyric Acid (GABA) Concentration | Baseline and at the end of each treatment cycle (each cycle is 21 days) during the treatment period.
  GABA levels in peripheral blood will be measured as an inhibitory neurotransmitter biomarker. Concentrations will be quantified using immunoassay or LC-MS.Unit of Measure: μmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Professor, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Upon completion of the study and following the publication of the paper, data supporting the findings of this study will be made available upon reasonable request from the Principal Investigator.